CLINICAL TRIAL: NCT06985771
Title: Evaluating the Predictive Ability of Different Frailty Indices for Postoperative Infections in Elderly Patients: Data Analysis From a Prospective Multicenter Observational Cohort
Brief Title: Predictive Ability of Different Frailty Indices for Postoperative Infections in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The First Medical Center of Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Deputy Chief Anesthesiologist, Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-L08
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Infections; Frailty
Keywords: Frailty; Postoperative Infection; elderly patients
MeSH Terms: conditions — Frailty | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative infection or not: Postoperative infection within 30 days postoperatively versus no infection.
  Interventions: Other: Observational study, with no intervention.

INTERVENTIONS:
Other: Observational study, with no intervention. — Observational study, with no intervention.

SUMMARY:
In this study, we extracted data from the patients medical record within the cohort to compare five existing frailty indices: the 5-Item Modified Frailty Index (mFI-5), the Electronic Frailty Index (eFI), the Frailty Index based on Comprehensive Geriatric Assessment (FI-CGA), the Frailty Risk Assessment Instrument for the Elderly based on Laboratory and Clinical Indicators (FRAIL), and the Hospital Frailty Risk Score (HFRS). The study aims to evaluate the predictive values of each electronic frailty index for the incidence of postoperative infection-related adverse events. This includes the primary outcome of infection events occurring within 30 days and the secondary outcome of the correlations among the five frailty indices.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 and above
2. Patients who underwent Non-Cardiac surgeries and anesthesia

Exclusion Criteria:

1. Patients who underwent surgery within 30 days before the current procedure;
2. Patients with missing baseline demographic data;
3. Patients with incomplete medical records that resulted in the inability to fully assess all five frailty indices;
4. Patients with missing data related to primary and secondary outcomes after surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The patients aged 65 and older who were involved in the prospective cohort of postoperative adverse events in elderly patients from April 2020 to April 2022.
Sampling Method: Non-Probability Sample
Enrollment: 10536 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Postoperative infection events within 30 days postoperatively | Within 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jingsheng Lou, Doctor, Principal Investigator — The First Medical Center of Chinese PLA General Hospital
Locations (1):
- The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided